CLINICAL TRIAL: NCT05242783
Title: The Effect of Intramyometrial Injection of Terlipressin Versus Carbitocin on Hemoglobin and Blood Loss During Open Myomectomy Operations Using Haemostatic Tourniquets: Double Blinded Randomized Placebo-Controlled Trial
Brief Title: The Effect of Intramyometrial Injection of Terlipressin Versus Carbitocin on Hemoglobin and Blood Loss During Open Myomectomy Operations Using Haemostatic Tourniquets:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wael Elbanna Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Elbanna_007
Record Dates: First submitted 2021-12-09; First posted 2022-02-16 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2022-02

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma | interventions — Terlipressin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects who meet diagnostic requirements as listed in the inclusion and exclusion criteria will be included in the study. Women will be randomized to one of the three arms using a computer-generated randomization table with a 1:1:1 group allocation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blinded randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- intramyometrial Terlipressin injection (Active Comparator): intramyometrial Terlipressin injection in women undergoing open myomectomy procedure using haemostatic tourniquets.
  (After the uterus has been reached, the Foley's urethral catheter will be adapted as a uterine tourniquet and will be applied at the base of the uterus before enucleating the fibroid masses. intramural Terlipressin will be injected, and then the uterine incision is done and the surgeon can now separate out the fibroids with ease and then amount of blood loss is calculated)
  Interventions: Drug: Terlipressin
- intramyometrial Carbetocin injection (Active Comparator): intramyometrial Carbetocin injection in women undergoing open myomectomy procedure using haemostatic tourniquets.
  (After the uterus has been reached, the Foley's urethral catheter will be adapted as a uterine tourniquet and will be applied at the base of the uterus before enucleating the fibroid masses. intramural carbitocin will be injected, and the uterine incision is done and the surgeon can now separate out the fibroids with ease and then amount of blood loss is calculated)
  Interventions: Drug: Terlipressin
- intramyometrial saline injection (Placebo Comparator): intramyometrial saline injection in women undergoing open myomectomy procedure using haemostatic tourniquets.
  After the uterus has been reached, the Foley's urethral catheter will be adapted as a uterine tourniquet and will be applied at the base of the uterus before enucleating the fibroid masses. intramural saline as a aplacebo will be injected, and the uterine incision is done and the surgeon can now separate out the fibroids with ease and then amount of blood loss is calculated) and amount of blood loss and operative time is compared between all arms
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — intramyometrial Terlipressin versus carbitocin versus saline(placebo) injection in women undergoing open myomectomy procedure using haemostatic tourniquets.
  Other Names: carbitocin; saline (placebo)

SUMMARY:
the study aims to evaluate the efficacy of intramyometrial Terlipressin injection versus intramyometrial Carbetocin injection on hemoglobin level in women undergoing abdominal myomectomy. Moreover, to evaluate their efficacy in decreasing blood loss on operative time and to describe the injection sequelae for the same population. This clinical study will be conducted in compliance with the clinical study protocol and applicable regulatory requirements.

DETAILED DESCRIPTION:
This study is a prospective, comparative, double-blinded randomized placebo-controlled trial and multi-center study that will be conducted at Wael ElBanna Clinic and the NRC site. The study participants' relevant medical records will be collected and reviewed after obtaining informed consent for the participants. Data will be pooled and presented in aggregate, without the identification of individual subjects.

The study materials that will be used will include blood tests and ultrasound. The study will involve three study arms:

* Arm 1: intramyometrial Terlipressin injection in women undergoing open myomectomy procedure using haemostatic tourniquets.
* Arm 2: intramyometrial Carbetocin injection in women undergoing open myomectomy procedure using haemostatic tourniquets.
* Arm 3: intramyometrial saline injection in women undergoing open myomectomy procedure using haemostatic tourniquets(placebo).

Subjects who meet diagnostic requirements as listed in the inclusion and exclusion criteria will be included in the study. Women will be randomized to one of the three arms using a computer-generated randomization table with a 1:1:1 group allocation

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 16-45 years
2. Appropriate medical status for open surgery (Largest Myoma size from 4 cm up to 20 cm)
3. Baseline hemoglobin ≥9 g/dl
4. No contra-indications to the use of glyopressin or carbitocin
5. Myoma-related symptoms, such as pelvic pressure or pain, menorrhagia, or infertility
6. Not pregnant at the time of presentation

Exclusion Criteria:

1. Previous myomectomy
2. History of bleeding disorders
3. Concurrent anticoagulation therapy
4. History of Uncontrolled ischaemic heart disease
5. Any pelvic abnormalities requiring concomitant surgery
6. Treatment with a GnRH agonist or ulipristal acetate within three months preceding surgery
7. Inability to understand and provide written informed consent.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women with fibroids undergo open myomectomy using hemostatic tournique
Enrollment: 99 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of intramyometrial Terlipressin injection versus intramyometrial Carbetocin injection in decreasing blood loss in women undergoing open myomectomy using haemostatic tourniquets. | 12 hours
  To evaluate the efficacy of intramyometrial Terlipressin injection versus intramyometrial Carbetocin injection in decreasing blood loss in women undergoing open myomectomy using haemostatic tourniquets( measuring the amount of blood loss in mm )

SECONDARY OUTCOMES:
1. To evaluate the efficacy of intramyometrial Terlipressin injection versus intramyometrial Carbetocin injection on hemoglobin level in women undergoing open myomectomy using haemostatic tourniquets. | 24 hours
  1. To evaluate the efficacy of intramyometrial Terlipressin injection versus intramyometrial Carbetocin injection on hemoglobin level in women undergoing open myomectomy using haemostatic tourniquets. ( to evaluate the change in hemoglobin level between before and after the operation )

CONTACTS AND LOCATIONS:
Locations (1):
- Wael El-Banna Clinic, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song T, Kim MK, Kim ML, Jung YW, Yun BS, Seong SJ. Use of vasopressin vs epinephrine to reduce haemorrhage during myomectomy: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2015 Dec;195:177-181. doi: 10.1016/j.ejogrb.2015.10.003. Epub 2015 Oct 24. PMID 26550945
- [Result] Parker WH, Berek JS, Pritts EA, Olive D, Chalas E, Clarke-Pearson D. Regarding "Incidence of Occult Uterine Malignancy Following Vaginal Hysterectomy with Morcellation". J Minim Invasive Gynecol. 2018 Sep-Oct;25(6):1113. doi: 10.1016/j.jmig.2018.04.008. Epub 2018 Apr 18. No abstract available. PMID 29679676
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21666469/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25767949/